CLINICAL TRIAL: NCT00174941
Title: Phase II, Open-Label Study, to Assess the Long-Term Safety of Oral TMX-67 in Subjects With Gout
Brief Title: Long-Term Safety of Febuxostat in Subjects With Gout.
Acronym: FOCUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMX-01-005; U1111-1114-2039 (Registry Identifier: WHO)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Gout
Keywords: Uric acid; xanthine oxidase; tophi; Drug Therapy
MeSH Terms: conditions — Gout | interventions — Febuxostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Febuxostat
- 2 (Experimental)
  Interventions: Drug: Febuxostat
- 3 (Experimental)
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Drug: Febuxostat — Febuxostat 40 mg, tablets, orally, once daily, based on serum urate level.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: 1
Drug: Febuxostat — Febuxostat 80 mg, tablets, orally, once daily, based on serum urate level.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: 2
Drug: Febuxostat — Febuxostat 120 mg, tablets, orally, once daily, based on serum urate level.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the long-term safety of febuxostat, once daily (QD), in maintaining serum urate levels within clinically acceptable levels in subjects with gout.

DETAILED DESCRIPTION:
Uric acid is the end product of purine degradation in humans. Hyperuricemia, a urate concentration in serum exceeding the limit of urate solubility (approximately 7.0 milligrams per deciliter [mg/dL]), is a common biochemical abnormality. Aberrations in any of the multiple mechanisms involved in the production and/or excretion of uric acid may increase serum urate concentrations, with persistent hyperuricemia as a marker for extracellular fluid monosodium urate supersaturation. As such, hyperuricemia is a necessary (but often not sufficient) risk factor for monosodium urate crystal deposition in tissues and is the fundamental pathophysiological process underlying the clinical manifestations of gout, which is a chronic disease characterized by urate crystal formation and deposition in joints and bones. Gout may progress from episodic attacks of acute inflammatory arthritis to a disabling chronic disorder characterized by deforming arthropathy; destructive deposits of urate crystals (tophi) in bones, joints, and other organs; structural and functional renal impairment due to interstitial urate crystal deposition; and urinary tract stones composed entirely or in part of uric acid crystals. Management of gout requires chronic treatment aimed at lowering serum urate into a subsaturating range (usually <6.0 mg/dL) in which crystal formation and deposition are prevented or reversed.

Febuxostat (TMX-67) is a non-purine selective xanthine oxidase inhibitor being developed as an orally administered agent for management of hyperuricemia in patients with gout.

Subjects who want to participate in this study will have successfully completed study TMX-00-004 (NCT00174967).

All participants will initially receive an 80 mg dose. Dose titrations will occur in order to obtain and maintain clinically acceptable serum urate levels.

ELIGIBILITY:
Inclusion Criteria:

* Hyperuricemia (serum uric acid ≥8.0 mg/dL upon entering parent study TMX-00-004).
* Must meet American College of Rheumatology criteria for gout.
* Must have adequate renal function (serum creatinine <1.5 mg/dL).
* Must have completed four weeks of double-blind dosing in Study TMX-00-004.
* Must not have experienced any serious study drug-related Adverse Events in Study TMX 00-004.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria:

* History of xanthinuria
* Alcohol consumption >14/week
* Has a History of significant concomitant illness
* Has active liver disease.
* Has a body mass index greater than 50 kg/m2
* Any other significant medical condition that would interfere with the treatment, safety or compliance with the protocol, as defined by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2001-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Takeda

REFERENCES:
- [Result] Colwell HH, Hunt BJ, Pasta DJ, Palo WA, Mathias SD, Joseph-Ridge N. Gout Assessment Questionnaire: Initial results of reliability, validity and responsiveness. Int J Clin Pract. 2006 Oct;60(10):1210-7. doi: 10.1111/j.1742-1241.2006.01104.x. Epub 2006 Aug 15. PMID 16911575
- [Result] Schumacher HR Jr, Becker MA, Lloyd E, MacDonald PA, Lademacher C. Febuxostat in the treatment of gout: 5-yr findings of the FOCUS efficacy and safety study. Rheumatology (Oxford). 2009 Feb;48(2):188-94. doi: 10.1093/rheumatology/ken457. PMID 19141576
- [Result] Whelton A, Macdonald PA, Zhao L, Hunt B, Gunawardhana L. Renal function in gout: long-term treatment effects of febuxostat. J Clin Rheumatol. 2011 Jan;17(1):7-13. doi: 10.1097/RHU.0b013e318204aab4. PMID 21169856
- See also: Uloric Package Insert — http://general.takedapharm.com/content/file.aspx?applicationcode=6C7C39D8-5D09-453B-BF30-696A4AB88E62&fileTypeCode=ULORICPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 23 investigational sites in the United States from 21 March 2001 to 29 December 2006
Pre-assignment Details: Subjects were to have completed 4 weeks of double-blind dosing in Study TMX-00-004 (NCT00174967) before enrollment in once daily (QD) treatment groups. Dose titrations will occur in order to obtain and maintain clinically acceptable serum urate levels.
Groups:
- Febuxostat 40 mg QD: Febuxostat 40 mg, orally, once daily, based on serum urate level.
- Febuxostat 80 mg QD: Febuxostat 80 mg, orally, once daily, based on serum urate level.
- Febuxostat 120 mg QD: Febuxostat 120 mg, orally, once daily, based on serum urate level.
Period: Overall Study
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Started | 8 (Subjects started on febuxostat 80mg. Number of subjects based on Final Stable Dose after titration.) | 79 (Subjects started on febuxostat 80mg. Number of subjects based on Final Stable Dose after titration.) | 29 (Subjects started on febuxostat 80mg. Number of subjects based on Final Stable Dose after titration.) | 116
Completed | 6 | 41 | 11 | 58
Not Completed | 2 | 38 | 18 | 58
Not completed — Adverse Event | 1 | 10 | 2 | 13
Not completed — Protocol Violation | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 3 | 2 | 5
Not completed — Personal Reason(s) | 0 | 14 | 8 | 22
Not completed — Gout Flare | 0 | 4 | 4 | 8
Not completed — Reason Not Specified | 1 | 6 | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Febuxostat 40 mg QD: Febuxostat 40 mg orally, once daily, based on serum urate level.
- Total: Total of all reporting groups
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total
Number analyzed (Participants) | 8 | 79 | 29 | 116
Age, Customized [Number; unit: Subjects]
  <45 years | 2 | 20 | 9 | 31
  45 to <65 years | 4 | 40 | 15 | 59
  ≥65 years | 2 | 19 | 5 | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 54.5 (11.44) | 53.9 (12.85) | 51.3 (13.01) | 53.3 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 9 | 2 | 11.0
  Male | 8 | 70 | 27 | 105.0
History of Kidney Stone [Number; unit: Subjects]
  Yes | 0 | 11 | 3 | 14
  No | 8 | 68 | 26 | 102
Presence of Tophus [Number; unit: Subjects]
  Yes | 1 | 13 | 12 | 26
  No | 7 | 66 | 17 | 90
Race/Ethnicity [Number; unit: Subjects]
  Asian | 0 | 0 | 2 | 2
  Black or African American | 1 | 5 | 3 | 9
  White | 7 | 71 | 21 | 99
  Hispanic | 0 | 2 | 1 | 3
  Other | 0 | 1 | 2 | 3
Renal Function [Number; unit: Subjects] — Impaired renal function was defined as serum creatinine >1.5 milligrams per deciliter (mg/dL) or a creatinine clearance of ≤80 milliliters per minute (mL/min)
  Subjects
    Normal | 3 | 33 | 12 | 48
    Impaired | 5 | 46 | 17 | 68
Urine Uric Acid [Number; unit: Subjects]
  Underexcretor | 5 | 62 | 21 | 88
  Overproducer | 3 | 16 | 7 | 26
  Missing | 0 | 1 | 1 | 2
Body Mass Index [Mean (Standard Deviation); unit: kiligram per meter² (kg/m²)] | 28.4 (2.78) | 32.9 (5.28) | 33.9 (6.82) | 32.9 (5.69)
Serum Urate [Mean (Standard Deviation); unit: mg/dL] | 9.58 (1.18) | 9.48 (1.04) | 10.23 (1.74) | 9.7 (1.30)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Whose Serum Urate Level Decreases to or is Maintained at <6.0 mg/dL at Month 6 Visit.
Description: Serum urate values were obtained at the Month 6 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Month 6 visit was summarized.
Time Frame: Month 6
Population: Subjects with a serum urate value at the Month 6 visit were included in the analysis. Results were summarized by the dose the subject was receiving at the Month 6 visit. Subjects must have been receiving that dose for at least 14 days prior to the visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 10 | 58 | 17 | 85
percentage of subjects | 50 | 93 | 65 | 82

2. Secondary Outcome: Percent Change in Serum Urate Levels From Baseline at Month 6 Visit.
Description: Serum urate values were obtained at the Month 6 visit. The percent change in serum urate from baseline to the Month 6 visit was summarized.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 10 | 58 | 17 | 85
percent change from baseline | -35.9 (9.55) | -50.6 (9.84) | -47.6 (19.6) | -48.3 (13.07)

3. Primary Outcome: Percentage of Subjects Whose Serum Urate Level Decreases to or is Maintained at <6.0 mg/dL at Month 12 Visit.
Description: Serum urate values were obtained at the Month 12 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Month 12 visit was summarized.
Time Frame: Month 12
Population: Subjects with a serum urate value at the Month 12 visit were included in the analysis. Results were summarized by the dose the subject was receiving at the Month 12 visit. Subjects must have been receiving that dose for at least 14 days prior to the visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 7 | 55 | 18 | 80
percentage of subjects | 57 | 85 | 67 | 79

4. Primary Outcome: Percentage of Subjects Whose Serum Urate Level Decreases to or is Maintained at <6.0 mg/dL at Month 18 Visit.
Description: Serum urate values were obtained at the Month 18 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Month 18 visit was summarized.
Time Frame: Month 18
Population: Subjects with a serum urate value at the Month 18 visit were included in the analysis. Results were summarized by the dose the subject was receiving at the Month 18 visit. Subjects must have been receiving that dose for at least 14 days prior to the visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 8 | 50 | 14 | 72
percentage of subjects | 50 | 82 | 57 | 74

5. Primary Outcome: Percentage of Subjects Whose Serum Urate Level Decreases to or is Maintained at <6.0 mg/dL at Month 24 Visit.
Description: Serum urate values were obtained at the Month 24 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Month 24 visit was summarized.
Time Frame: Month 24
Population: Subjects with a serum urate value at the Month 24 visit were included in the analysis. Results were summarized by the dose the subject was receiving at the Month 24 visit. Subjects must have been receiving that dose for at least 14 days prior to the visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 8 | 49 | 13 | 70
percentage of subjects | 63 | 76 | 92 | 77

6. Primary Outcome: Percentage of Subjects Whose Serum Urate Level Decreases to or is Maintained at <6.0 mg/dL at Month 36 Visit.
Description: Serum urate values were obtained at the Month 36 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Month 36 visit was summarized.
Time Frame: Month 36
Population: Subjects with a serum urate value at the Month 36 visit were included in the analysis. Results were summarized by the dose the subject was receiving at the Month 36 visit. Subjects must have been receiving that dose for at least 14 days prior to the visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 6 | 45 | 13 | 64
percentage of subjects | 67 | 84 | 92 | 84

7. Primary Outcome: Percentage of Subjects Whose Serum Urate Level Decreases to or is Maintained at <6.0 mg/dL at Month 48 Visit.
Description: Serum urate values were obtained at the Month 48 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Month 48 visit was summarized.
Time Frame: Month 48
Population: Subjects with a serum urate value at the Month 48 visit were included in the analysis. Results were summarized by the dose the subject was receiving at the Month 48 visit. Subjects must have been receiving that dose for at least 14 days prior to the visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 6 | 39 | 13 | 58
percentage of subjects | 83 | 92 | 85 | 90

8. Primary Outcome: Percentage of Subjects Whose Serum Urate Level Decreases to or is Maintained at <6.0 mg/dL at Month 60 Visit.
Description: Serum urate values were obtained at the Month 60 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Month 60 visit was summarized.
Time Frame: Month 60
Population: Subjects with a serum urate value at the Month 60 visit were included in the analysis. Results were summarized by the dose the subject was receiving at the Month 60 visit. Subjects must have been receiving that dose for at least 14 days prior to the visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 6 | 41 | 11 | 58
percentage of subjects | 100 | 93 | 91 | 93

9. Primary Outcome: Percentage of Subjects Whose Serum Urate Level Decreases to or is Maintained at <6.0 mg/dL at Final Visit.
Description: The percentage of subjects whose serum urate was <6.0 mg/dL at the final visit was summarized. The final visit was the last visit at which a serum urate value was collected.
Time Frame: Last Visit on treatment (up to 66 months).
Population: Two subjects who did not have any post-baseline Serum Urate Level measurements were excluded from this analysis. Results were summarized by the dose the subject was receiving at the time of the final visit. Subjects must have been receiving that dose for at least 14 days prior to the visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 8 | 79 | 27 | 114
percentage of subjects | 100 | 82 | 81 | 83

10. Secondary Outcome: Percent Change in Serum Urate Levels From Baseline at Month 12 Visit.
Description: Serum urate values were obtained at the Month 12 visit. The percent change in serum urate from baseline to the Month 12 visit was summarized.
Time Frame: Baseline and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 7 | 55 | 18 | 80
percentage of subjects | -35.0 (13.16) | -49.7 (9.26) | -49.3 (15.77) | -48.3 (11.94)

11. Secondary Outcome: Percent Change in Serum Urate Levels From Baseline at Month 18 Visit.
Description: Serum urate values were obtained at the Month 18 visit. The percent change in serum urate from baseline to the Month 18 visit was summarized.
Time Frame: Baseline and Month 18
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 8 | 50 | 14 | 72
percent change from baseline | -35.5 (16.35) | -48.7 (11.12) | -39.5 (19.36) | -45.4 (14.35)

12. Secondary Outcome: Percent Change in Serum Urate Levels From Baseline at Month 24 Visit.
Description: Serum urate values were obtained at the Month 24 visit. The percent change in serum urate from baseline to the Month 24 visit was summarized.
Time Frame: Baseline and Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 8 | 49 | 13 | 70
percent change from baseline | -38.9 (19.41) | -46.7 (11.59) | -54.7 (12.02) | -47.3 (13.24)

13. Secondary Outcome: Percent Change in Serum Urate Levels From Baseline at Month 36 Visit.
Description: Serum urate values were obtained at the Month 36 visit. The percent change in serum urate from baseline to the Month 36 visit was summarized.
Time Frame: Baseline and Month 36
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 6 | 45 | 13 | 64
percent change from baseline | -43.0 (9.14) | -46.9 (13.35) | -56.4 (13.76) | -48.4 (13.6)

14. Secondary Outcome: Percent Change in Serum Urate Levels From Baseline at Month 48 Visit.
Description: Serum urate values were obtained at the Month 48 visit. The percent change in serum urate from baseline to the Month 48 visit was summarized.
Time Frame: Baseline and Month 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 6 | 39 | 13 | 58
percent change from baseline | -50.0 (4.16) | -50.3 (10.61) | -53.8 (16.41) | -51.1 (11.64)

15. Secondary Outcome: Percent Change in Serum Urate Levels From Baseline at Month 60 Visit.
Description: The secondary outcome was the mean percent change from baseline to Month 60 visit as assessed by serum urate levels collected at baseline and at the Month 60 visit by dose at observation.
Time Frame: Baseline and Month 60
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 6 | 41 | 11 | 58
percent change from baseline | -45.5 (8.70) | -51.1 (13.21) | -59.0 (18.74) | -52.0 (14.32)

16. Secondary Outcome: Percent Change in Serum Urate Levels From Baseline at Final Visit.
Description: The percent change in serum urate from baseline to the final visit was summarized. The final visit was the last visit at which a serum urate value was collected.
Time Frame: Baseline and Last Visit on treatment (up to 66 months).
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Total Febuxostat
Number analyzed (Participants) | 8 | 79 | 27 | 114
percent change from baseline | -49.2 (7.10) | -47.1 (16.42) | -50.7 (19.12) | -48.1 (16.61)

ADVERSE EVENTS:
Groups:
- Febuxostat 40 mg QD: Febuxostat 40 mg taken orally, once daily, based on serum urate level.
- Febuxostat 80 mg QD: Febuxostat 80 mg, taken orally, once daily, based on serum urate level
- Febuxostat 120 mg QD: Febuxostat 120 mg, taken orally, once daily, based on serum urate level
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Febuxostat Total
Serious Adverse Events (participants affected / at risk) | 3/12 | 14/116 | 4/37 | 21/116
Other Adverse Events (participants affected / at risk) | 5/12 | 44/116 | 9/37 | 53/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat 40 mg QD (N=12) | Febuxostat 80 mg QD (N=116) | Febuxostat 120 mg QD (N=37) | Febuxostat Total (N=116)
Cardiac Conduction Disorders (Cardiac disorders) | 0 | 1 | 0 | 1
Supraventricular Arrhythmias (Cardiac disorders) | 0 | 5 | 0 | 5
Duodenal and Small Intestinal Stenosis and Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal Ulcers and Perforation, Site Unspecified (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Intestinal Ulcers & Perforation not elsewhere classified (NEC) (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pain and Discomfort NEC (General disorders) | 0 | 1 | 0 | 1
Cholecystitis and Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | 2
Abdominal and Gastrointestinal Infections (Infections and infestations) | 0 | 1 | 0 | 1
Lower Respiratory Tract and Lung Infections (Infections and infestations) | 1 | 1 | 0 | 2
Sepsis, Bacteraemia, Viraemia, and Infections (Infections and infestations) | 0 | 1 | 0 | 1
Cerebral Injuries NEC (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Fractures and Dislocations NEC (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Non-Site Specific Injuries NEC (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Radiation Injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Intervertebral Disc Disorders (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Joint Related Disorders NEC (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteoarthropathies (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Pathological Fractures and Complications (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Spine and Neck Deformities (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Lip and Oral Cavity Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Prostatic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Respiratory Tract and Pleural Neoplasms Benign NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Skin Neoplasms Malignant & Unspecified (Excluding Melanoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Alzheimer's Disease (Including Subtypes) (Nervous system disorders) | 0 | 1 | 0 | 1
Central Nervous System Hemorrhages & Cerebrovascular Accidents (Nervous system disorders) | 1 | 0 | 0 | 1
Depressive Disorders (Psychiatric disorders) | 1 | 0 | 0 | 1
Bladder and Urethral Symptoms (Renal and urinary disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat 40 mg QD (N=12) | Febuxostat 80 mg QD (N=116) | Febuxostat 120 mg QD (N=37) | Febuxostat Total (N=116)
Diarrhoea (Gastrointestinal disorders) | 0 | 9 | 1 | 10
Liver Function Analyses (Investigations) | 0 | 4 | 2 | 6
Gastrointestinal Atonic and Hypomotility Disorders NEC (Gastrointestinal disorders) | 0 | 5 | 0 | 5
Headaches NEC (Nervous system disorders) | 0 | 5 | 0 | 5
Hyperlipidaemias NEC (Metabolism and nutrition disorders) | 1 | 3 | 0 | 4
White Blood Cell Analyses (Investigations) | 0 | 3 | 0 | 3
Muscle Related Signs and Symptoms NEC (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 3
Renal Lithiasis (Renal and urinary disorders) | 1 | 2 | 0 | 3
Rashes, Eruptions and Exanthems (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 3
Gastrointestinal Signs and Symptoms (Gastrointestinal disorders) | 0 | 3 | 1 | 3
Nausea and Vomiting Symptoms (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Oedema NEC (General disorders) | 0 | 2 | 0 | 2
Triglyceride Analyses (Investigations) | 0 | 2 | 0 | 2
Arthropathies (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Joint Related Signs and Symptoms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Muscle Pains (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Musculoskeletal and Connective Tissue Signs and Symptoms NEC (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Blood Amylase Increased (Investigations) | 1 | 0 | 0 | 1
Skin Injuries NEC (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Weight Increased (Investigations) | 0 | 0 | 1 | 1
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.